CLINICAL TRIAL: NCT01845948
Title: Effectiveness of a Parental Training Programme to Enhance Parent-child Relationship and Reduce Harsh Parenting Practices and Parental Stress in the Preparation of Children for Transition to Primary School: A Randomized Controlled Trial
Brief Title: Effectiveness of a Parental Training Programme to Enhance Parent-child Relationship and Reduce Harsh Parenting Practices and Parental Stress in the Preparation of Children for Transition to Primary School
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. LI William Ho Cheung, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ND789
Record Dates: First submitted 2013-04-25; First posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Parent
Keywords: parents; school transition; parental-child relationship

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Control (Placebo Comparator): Parents had no intervention except that an information leaflet for parents on helping children to adapt the new primary school life published by Education Bureau was given to each parent in the control group at the end of data collection.
  Interventions: Behavioral: Placebo Control
- parental training programme (Experimental): The parental training programme was run in small groups of 8 to 12 parents over four consecutive weeks. They consisted of four group sessions, each lasting about two hours. The major focus of the parental intervention included teaching parents: (1) to use more active listening skills, (2) to engage less in harsh parenting practices, (3) to use more praise and encouragement and (4) to set reasonable expectations in the rearing of their children. Each session was started with revision of skills or concepts discussed in previous sessions, therefore, each session built on the previous session.
  Interventions: Behavioral: parental training programme

INTERVENTIONS:
Behavioral: parental training programme — In the experimental group, parents participated in the parental training programme approximately one month before the start of the academic year in primary school. Two social workers, who have minimum five- year experience in giving family counselling,implemented the interventions.
  Arms: parental training programme
Behavioral: Placebo Control — Parents had no intervention except that an information leaflet for parents on helping children to adapt the new primary school life published by Education Bureau was given to each parent in the control group at the end of data collection.
  Arms: Placebo Control

SUMMARY:
This study tested the effectiveness of a parental training programme to enhance parent-child relationship and reduce harsh parenting practices and parental stress in the preparation of children for transition to primary school. A randomized controlled trial was employed and 142 parents were recruited. Parents in the experimental group engaged in less harsh parenting practices and reported better parent-child relationships than parents in the control group. Findings from this study provide empirical evidence of the effectiveness of the parental training programme and highlight the significance of parental involvement in promoting a smooth transition for children from kindergarten to primary one.

DETAILED DESCRIPTION:
Introduction Transition creates a time of vulnerability for the child, the parents and their relationship. Failure to adjust to the transition, on the part of either parents or children, might place the family in a psychological devastating position. There is an imperative need to develop and evaluate appropriate interventions for parents so that they can contribute to helping their children enjoy a smooth passage to a pleasurable learning life in primary school.

Aim The aims of this study were to test the effectiveness of a parental training programme to enhance parent-child relationship and reduce harsh parenting practices and parental stress in the preparation of children for transition to primary school.

Methods A randomized controlled trial, two-group pre-test and repeated post-test, between-subjects design was employed. The method of simple complete randomization was adopted. Recruitment and data collection were conducted during the summer in 2009. Participants were recruited through referrals from the Hong Kong Sheung Kung Hui Welfare Council in Tung Chung. Written consent was obtained from parents after they were told the purposes of the study and agreed to participate. Parents were told that they were under no obligation to participate, could withdraw from the study with impunity at any time and were assured of the confidentiality of the data to be collected.

After they had signed consent forms, a research assistant collected demographic and baseline data from parents. Data collection was divided into three phases: at the time of recruitment (pre-intervention), at six weeks and three months after the intervention. Parents were asked to respond to the Chinese version of the parental acceptance-rejection scale, parental stress scale, and self-report scale on parent-child relationship in respect of the transition from kindergarten to primary school.

ELIGIBILITY:
Inclusion Criteria:

* must be able to read and write Chinese
* must have had primary school education or above

Exclusion Criteria:

* with identified cognitive and learning problems were excluded, as also were children with such problems

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change of Self-reported Parent-Child Relationship at 6 weeks from baseline | 6 weeks
  The parent-child relationship of the participants was measured by using a self-reporting method consisting of two items, with one asking 'How satisfied are you with the parent-child relationship?" and the other 'As a parent, how satisfied are you with yourself?'

SECONDARY OUTCOMES:
Self-reported Parent-Child Relationship at baseline | baseline, 0 week ( just before the start of intervention)
  The parent-child relationship of the participants was measured by using a self-reporting method consisting of two items, with one asking 'How satisfied are you with the parent-child relationship?" and the other 'As a parent, how satisfied are you with yourself?'
Change of Self-reported Parent-Child Relationship at 3 months from baseline | 3 months
  The parent-child relationship of the participants was measured by using a self-reporting method consisting of two items, with one asking 'How satisfied are you with the parent-child relationship?" and the other 'As a parent, how satisfied are you with yourself?'
Perceived Parental Aggression Scale at baseline | baseline, 0 week ( just before the start of intervention)
  It measures harsh parenting, i.e. physical or verbal aggression towards children
change of Perceived Parental Aggression Scale at 6 weeks from baseline | 6 weeks
  It measures harsh parenting, i.e. physical or verbal aggression towards children
change of Perceived Parental Aggression Scale at 3 months from baseline | 3 months
  It measures harsh parenting, i.e. physical or verbal aggression towards children
Parental Stress at baseline | baseline, 0 week ( just before the start of intervention)
  we assess a parent's subjective feelings of strain, difficulty and dissatisfaction in reaction to stressors in the parent-child relationship
change of Parental Stress at baseline at 6 weeks from baseline | 6 weeks
  we assess a parent's subjective feelings of strain, difficulty and dissatisfaction in reaction to stressors in the parent-child relationship
change of Parental Stress at baseline at 3 months from baseline | 3 months
  we assess a parent's subjective feelings of strain, difficulty and dissatisfaction in reaction to stressors in the parent-child relationship

CONTACTS AND LOCATIONS:
Overall Officials: William Ho Cheung Li, PhD, Principal Investigator — The School of Nursing, The University of Hong Kong
Locations (1):
- Hong Kong Sheng Kung Hui Tung Chung Integrated Services, Hong Kong, China

REFERENCES:
- [Derived] Li HC, Chan SS, Mak YW, Lam TH. Effectiveness of a parental training programme in enhancing the parent-child relationship and reducing harsh parenting practices and parental stress in preparing children for their transition to primary school: a randomised controlled trial. BMC Public Health. 2013 Nov 16;13:1079. doi: 10.1186/1471-2458-13-1079. PMID 24237718